CLINICAL TRIAL: NCT04885231
Title: Impact of Counseling and Education on Opioid Consumption After Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Trial
Brief Title: Impact of Counseling and Education on Opioid Consumption After ACL Reconstruction
Acronym: CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Jonathan D. Packer, MD, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00093883
Record Dates: First submitted 2021-05-02; First posted 2021-05-13 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Pain, Postoperative; Opioid Use
MeSH Terms: conditions — Pain, Postoperative | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: Single center randomized control trial consisting of two groups - one control and one experimental.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid-Limiting Perioperative Pain Management Education and Counseling (Experimental): Patients will be instructed to take oxycodone only as a last resort if the pain becomes unbearable. "The goal should be to take as little oxycodone as possible."
  Interventions: Behavioral: Perioperative Pain Management Education and Counseling
- Traditional Perioperative Pain Management Education and Counseling (Active Comparator): Patients will be instructed to take opioids as needed for severe pain to manage and "stay ahead" of the postoperative pain
  Interventions: Behavioral: Perioperative Pain Management Education and Counseling

INTERVENTIONS:
Behavioral: Perioperative Pain Management Education and Counseling — All patients will receive both verbal postoperative pain management education and counseling as well as a written handout. Multi-modality non-opioid methods of pain control will be thoroughly discussed.

SUMMARY:
Research question: Does an opioid limiting pain management counseling and education program result in decreased opioid consumption and improved pain control compared to traditional pain management programs after anterior cruciate ligament reconstruction (ACLR) surgery?

At many institutions, the current standard of care is to instruct patients to take opioid pain medicine as needed when in severe pain to "stay ahead of the pain." This study is investigating whether modifying the instructions to take opioid pain medications only if in "unbearable pain" will have an effect on 1) reducing opioid consumption and 2) improving pain levels.

Adults who are undergoing an ACLR surgery will be invited to participate in the study and be randomly assigned to one of the two pain management programs. All patients will receive a comprehensive multi-modality pain management treatments and medications. Patients in both groups will receive the same type and amount of all postoperative medications. The only difference will be in the instructions about when to take the opioid medications.

The patients will then be sent an electronic survey twice per day for 2 weeks about their pain levels and number of opioid pills taken.

DETAILED DESCRIPTION:
Prescription narcotic pain medications (opioids) were responsible for roughly 17,000 deaths in 2016 in the United States. Orthopedic surgeons were responsible for prescribing the third highest percentage of opioids among physicians in 2009. In recent years, orthopaedic surgeons have used many different types of non-opioid pain medications and methods to reduce patients' opioid after surgery. Opioid dependence can manifest from prescription use, especially in patients who have never used opioids before.

The purpose of this study is to research the effect of different pain management education programs on pain control and opioid use after an anterior cruciate ligament reconstruction (ACLR) surgery. Specifically, does education directed at avoiding opioids unless in "unbearable pain" have any effect on reducing pain levels and opioid consumption in the early postoperative period compared to traditional pain management education?

Patients who agree to participate in this study will be assigned at random to two opioid education programs after ACLR. All patients will be given peri-operative pain management counseling and education. Patients in the experimental group will be instructed to avoid opioids unless in unbearable pain. Patients in the control group will be instructed to take opioid medication as needed for severe pain to "stay ahead" of the pain. Participants in both groups will be prescribed the exact same type and amount of postoperative medications.

Surveys will be sent electronically to patients twice per day for 2 weeks to monitor pain levels and the amount of opioid consumption. Also, patients will be asked to complete demographic and patient-reported outcome questionnaires after surgery. Patients will be involved in the study for 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 14 years and older
2. All patients scheduled to undergo an ACLR with or without concomitant procedures such as arthroscopic cartilage procedures, meniscus repair or meniscectomy, and/or lateral extraarticular tenodesis (anterolateral ligament reconstruction)
3. Willing to participate in a perioperative pain management education and counseling program
4. Willing to track pain levels and opioid consumption through surveys administered via text
5. Willing to receive a perioperative regional nerve block
6. Language skills and cognitive ability required to participate in the study
7. Provision of informed consent

Exclusion Criteria:

1. Revision ACLR
2. Concomitant open cartilage procedures or additional knee ligament repair or reconstruction
3. Concomitant injury that would also influence pain management
4. History of heroin use or opioid abuse requiring treatment
5. If any previous ipsilateral knee surgery except for knee arthroscopy
6. Preoperative Kellgren-Lawrence grade 3 and 4 on weightbearing radiographs
7. An allergy to any of the study medications
8. Previously enrolled in the CARE trial
9. Anticipated problems with the patient returning for follow-up or accurate completion of survey
10. If patient cannot reliably receive texts and use internet to complete surveys

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 3 months
  The total morphine equivalents (TMEs) consumed by the patient after surgery

SECONDARY OUTCOMES:
Numeric Pain Scale | Two weeks
  Participants will record a Numeric Pain Scale (NPS) score every day on a scale of 0-10, where 0= no pain and 10= worst possible pain. Mean NPS values for each postoperative day will be compared between groups.
Patient Reported Outcomes - Satisfaction with social roles & activities | 2 weeks, 6 weeks, 3 months
  Patient reported social satisfaction will be assessed after surgery using PROMIS Satisfaction with Social roles and Activities questionnaire
Patient Reported Outcomes - Physical Function | 2 weeks, 6 weeks, 3 months
  Patient reported physical functioning will be assessed after surgery using PROMIS Physical Function questionnaire
Patient Reported Outcomes - Pain | 2 weeks, 6 weeks, 3 months
  Patient reported pain will be assessed after surgery using PROMIS Pain Interference questionnaire
Patient Reported Outcomes - Fatigue | 2 weeks, 6 weeks, 3 months
  Patient reported fatigue will be assessed after surgery using PROMIS Fatigue questionnaire
Patient Reported Outcomes - Depression | 2 weeks, 6 weeks, 3 months
  Patient reported depression will be assessed after surgery using PROMIS Emotional Distress - Depression questionnaire
Patient Reported Outcomes - Anxiety | 2 weeks, 6 weeks, 3 months
  Patient reported anxiety will be assessed after surgery using PROMIS Emotional Distress - Anxiety questionnaire
Opioid Prescription Refills | 3 months
  The mean number of opioid prescription refills per patient will be compared between the two treatment groups.
Patient Satisfaction | 2 weeks, 6 weeks, and 3 months
  Patient satisfaction will be assessed by the Surgical Satisfaction Survey (SSQ-8), with responses ranging from Very Satisfied to Very Unsatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D. Packer, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Rehabilitation and Orthopaedic Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borovkov SA, Shevchuk AG. [Rheologic properties of blood in chronic ischemia of the lower extremities]. Khirurgiia (Mosk). 1982 Jul;(7):44-7. No abstract available. Russian. PMID 7120832
- [Background] Aso K, Izumi M, Sugimura N, Okanoue Y, Kamimoto Y, Yokoyama M, Ikeuchi M. Additional benefit of local infiltration of analgesia to femoral nerve block in total knee arthroplasty: double-blind randomized control study. Knee Surg Sports Traumatol Arthrosc. 2019 Jul;27(7):2368-2374. doi: 10.1007/s00167-018-5322-7. Epub 2018 Dec 8. PMID 30536047
- [Background] Dysart SH, Barrington JW, Del Gaizo DJ, Sodhi N, Mont MA. Local Infiltration Analgesia With Liposomal Bupivacaine Improves Early Outcomes After Total Knee Arthroplasty: 24-Hour Data From the PILLAR Study. J Arthroplasty. 2019 May;34(5):882-886.e1. doi: 10.1016/j.arth.2018.12.026. Epub 2018 Dec 25. PMID 30799269
- [Background] Hyland SJ, Deliberato DG, Fada RA, Romanelli MJ, Collins CL, Wasielewski RC. Liposomal Bupivacaine Versus Standard Periarticular Injection in Total Knee Arthroplasty With Regional Anesthesia: A Prospective Randomized Controlled Trial. J Arthroplasty. 2019 Mar;34(3):488-494. doi: 10.1016/j.arth.2018.11.026. Epub 2018 Nov 23. PMID 30554925
- [Background] Kim N, Matzon JL, Abboudi J, Jones C, Kirkpatrick W, Leinberry CF, Liss FE, Lutsky KF, Wang ML, Maltenfort M, Ilyas AM. A Prospective Evaluation of Opioid Utilization After Upper-Extremity Surgical Procedures: Identifying Consumption Patterns and Determining Prescribing Guidelines. J Bone Joint Surg Am. 2016 Oct 19;98(20):e89. doi: 10.2106/JBJS.15.00614. PMID 27869630
- [Background] Kuang MJ, Du Y, Ma JX, He W, Fu L, Ma XL. The Efficacy of Liposomal Bupivacaine Using Periarticular Injection in Total Knee Arthroplasty: A Systematic Review and Meta-Analysis. J Arthroplasty. 2017 Apr;32(4):1395-1402. doi: 10.1016/j.arth.2016.12.025. Epub 2016 Dec 23. PMID 28082044
- [Background] Kumar K, Gulotta LV, Dines JS, Allen AA, Cheng J, Fields KG, YaDeau JT, Wu CL. Unused Opioid Pills After Outpatient Shoulder Surgeries Given Current Perioperative Prescribing Habits. Am J Sports Med. 2017 Mar;45(3):636-641. doi: 10.1177/0363546517693665. Epub 2017 Feb 9. PMID 28182507
- [Background] Kunze KN, Polce EM, Lilly DT, Garcia FL, Cohn MR, Nho SJ, Chahla J. Adjunct Analgesia Reduces Pain and Opioid Consumption After Hip Arthroscopy: A Systematic Review of Randomized Controlled Trials. Am J Sports Med. 2020 Dec;48(14):3638-3651. doi: 10.1177/0363546520905884. Epub 2020 Mar 2. PMID 32119562
- [Background] McLaughlin DC, Cheah JW, Aleshi P, Zhang AL, Ma CB, Feeley BT. Multimodal analgesia decreases opioid consumption after shoulder arthroplasty: a prospective cohort study. J Shoulder Elbow Surg. 2018 Apr;27(4):686-691. doi: 10.1016/j.jse.2017.11.015. Epub 2018 Jan 3. PMID 29305103
- [Background] Namdari S, Nicholson T, Abboud J, Lazarus M, Steinberg D, Williams G. Interscalene Block with and without Intraoperative Local Infiltration with Liposomal Bupivacaine in Shoulder Arthroplasty: A Randomized Controlled Trial. J Bone Joint Surg Am. 2018 Aug 15;100(16):1373-1378. doi: 10.2106/JBJS.17.01416. PMID 30106818
- [Background] Pitchon DN, Dayan AC, Schwenk ES, Baratta JL, Viscusi ER. Updates on Multimodal Analgesia for Orthopedic Surgery. Anesthesiol Clin. 2018 Sep;36(3):361-373. doi: 10.1016/j.anclin.2018.05.001. Epub 2018 Jul 11. PMID 30092934
- [Background] Rucinski K, Cook JL. Effects of preoperative opioid education on postoperative opioid use and pain management in orthopaedics: A systematic review. J Orthop. 2020 Jan 21;20:154-159. doi: 10.1016/j.jor.2020.01.020. eCollection 2020 Jul-Aug. PMID 32025140
- [Background] Schoenfeld AJ, Jiang W, Chaudhary MA, Scully RE, Koehlmoos T, Haider AH. Sustained Prescription Opioid Use Among Previously Opioid-Naive Patients Insured Through TRICARE (2006-2014). JAMA Surg. 2017 Dec 1;152(12):1175-1176. doi: 10.1001/jamasurg.2017.2628. PMID 28813584
- [Background] Sethi PM, Brameier DT, Mandava NK, Miller SR. Liposomal bupivacaine reduces opiate consumption after rotator cuff repair in a randomized controlled trial. J Shoulder Elbow Surg. 2019 May;28(5):819-827. doi: 10.1016/j.jse.2019.01.008. Epub 2019 Mar 28. PMID 30928396
- [Background] Sun EC, Darnall BD, Baker LC, Mackey S. Incidence of and Risk Factors for Chronic Opioid Use Among Opioid-Naive Patients in the Postoperative Period. JAMA Intern Med. 2016 Sep 1;176(9):1286-93. doi: 10.1001/jamainternmed.2016.3298. PMID 27400458
- [Background] Syed UAM, Aleem AW, Wowkanech C, Weekes D, Freedman M, Tjoumakaris F, Abboud JA, Austin LS. Neer Award 2018: the effect of preoperative education on opioid consumption in patients undergoing arthroscopic rotator cuff repair: a prospective, randomized clinical trial. J Shoulder Elbow Surg. 2018 Jun;27(6):962-967. doi: 10.1016/j.jse.2018.02.039. Epub 2018 Mar 26. PMID 29599038
- [Background] Tedesco D, Gori D, Desai KR, Asch S, Carroll IR, Curtin C, McDonald KM, Fantini MP, Hernandez-Boussard T. Drug-Free Interventions to Reduce Pain or Opioid Consumption After Total Knee Arthroplasty: A Systematic Review and Meta-analysis. JAMA Surg. 2017 Oct 18;152(10):e172872. doi: 10.1001/jamasurg.2017.2872. Epub 2017 Oct 18. PMID 28813550
- [Background] Volkow ND, McLellan TA, Cotto JH, Karithanom M, Weiss SR. Characteristics of opioid prescriptions in 2009. JAMA. 2011 Apr 6;305(13):1299-301. doi: 10.1001/jama.2011.401. No abstract available. PMID 21467282
- [Background] Xiao K, Yu L, Xiao W, Peng H, Bian Y, Wu Z, Weng X. Pain Management Using Perioperative Administration of Parecoxib for Total Hip Arthroplasty: A Randomized, Double-Blind, Placebo-Controlled Trial. Pain Physician. 2019 Nov;22(6):575-582. PMID 31775404